CLINICAL TRIAL: NCT06687538
Title: The Effect of Education to be Provided to Patients to Undergo Prostate Surgery With Mobile Application on Patient Outcomes
Brief Title: Effect of Education to be Provided to Patients to Undergo TURP With Mobile Application on Patient Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other); Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TU-BOZKUL-010
Record Dates: First submitted 2024-11-09; First posted 2024-11-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: Mobile application; Patient education; Patient outcomes; Nursing; Transurethral prostate resection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm (1:1), randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the data collection process, when the patients were admitted to the urology clinic, their inclusion in the study will be evaluated by the consultant M.B. and the executive G.B. Patients who meet the inclusion criteria will be assigned to the control and mobile application arm by block randomization (1:1) according to permutations (BABBAB, AABBAB) created in the computer environment by a statistical expert not involved in the study. After the randomization list is created, which letter (A, B) will represent which group will be determined by lottery method. The other consultant (SY), who will not be involved in the data collection process of the research, will write numbers from 1 to 68 on the envelopes as many as the number of the sample and letters representing the groups according to the randomization list will be added to each envelope. When a patient meets the inclusion criteria, agrees to participate in the study and signs the informed consent form, the GB will inform the co
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application group (Experimental): When the executive (EP) goes to the patient for the procedure, he/she will fill out the "Informed Consent Form", open the envelope and find out which group the patient is in. "Introductory Information Form", 'State Anxiety Scale', 'Hemodynamic Variables Monitoring Form' and 'Surgical Fear Scale' will be completed for all patients undergoing TURP. Patients in the study group will be introduced to the training to be given with the mobile application and downloaded to their phones/tablets. According to randomization, patients in the study group will receive training with the mobile application and patients in the control group will receive routine care. In the postoperative period, "Hemodynamic Variables Monitoring Form", "Visual Analog Scale" and "Discharge Training Satisfaction Scale" will be completed for all patients.
  Interventions: Other: Mobile application
- Control group (No Intervention): When the executive (EP) goes to the patient for the procedure, he/she will fill out the "Informed Consent Form", open the envelope and find out which group the patient is in. "Introductory Information Form", 'State Anxiety Scale', 'Hemodynamic Variables Monitoring Form' and 'Surgical Fear Scale' will be filled out for all patients who will undergo TURP. Patients in the control group will receive routine care. In the postoperative period, "Hemodynamic Variables Monitoring Form", "Visual Analog Scale" and "Discharge Training Satisfaction Scale" will be completed for all patients.

INTERVENTIONS:
Other: Mobile application — The content of the mobile application training to be developed for patients who will undergo transurethral prostate resection will consist of 3 modules including preoperative, postoperative and discharge training process.
  Arms: Mobile application group

SUMMARY:
The aim of this study was to determine the effect of mobile application training on patient outcomes (preoperative anxiety, surgical fear, postoperative pain, hemodynamic parameters, satisfaction level and length of hospital stay) in patients undergoing transurethral prostate resection surgery. It was planned as a prospective, two-arm (1:1), randomized controlled clinical trial. The study will be conducted with 68 patients in the urology clinic of a vir university hospital. Patients will be randomly assigned to the control group and the mobile application training group. Patients in the mobile application group will be trained with the mobile application, while patients in the control group will only receive routine care in the clinic. Patients assigned to the mobile application group will be introduced to the education to be given with the mobile application and the application will be downloaded to their phones/tablets. Data will be collected with the Introductory Information Form, Visual Comparison Scale, State Anxiety Scale, Hemodynamic Parameters Monitoring Form, Surgical Fear Scale and Discharge Education Satisfaction Scale. When the patient is admitted to the clinic, "Introductory Information Form", "State Anxiety Scale", and "Surgical Fear Scale" will be applied to the patients in the mobile intervention and control groups before surgical intervention, and "Hemodynamic Parameters Monitoring Form" will be completed. After the surgical intervention, "Visual Comparison Scale" and "Discharge Education Satisfaction Scale" will be applied to all patients and "Hemodynamic Parameters Monitoring Form" will be completed. The data will be analyzed in a computer environment.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of mobile application training on patient outcomes (preoperative anxiety, surgical fear, postoperative pain, hemodynamic parameters, satisfaction level and length of hospital stay) in patients undergoing transurethral prostate resection surgery. It was planned as a prospective, two-arm (1:1), randomized controlled clinical trial. The study will be conducted with 68 patients in the urology clinic of a vir university hospital. Patients will be randomly assigned to the control group and the mobile application training group. Patients in the mobile application group will be trained with the mobile application, while patients in the control group will only receive routine care in the clinic. Patients assigned to the mobile application group will be introduced to the education to be given with the mobile application and the application will be downloaded to their phones/tablets. Data will be collected with the Introductory Information Form, Visual Comparison Scale, State Anxiety Scale, Hemodynamic Parameters Monitoring Form, Surgical Fear Scale and Discharge Education Satisfaction Scale. When the patient is admitted to the clinic, "Introductory Information Form", "State Anxiety Scale", and "Surgical Fear Scale" will be applied to the patients in the mobile intervention and control groups before surgical intervention, and "Hemodynamic Parameters Monitoring Form" will be completed. After the surgical intervention, "Visual Comparison Scale" and "Discharge Education Satisfaction Scale" will be applied to all patients and "Hemodynamic Parameters Monitoring Form" will be completed. The data will be analyzed in a computer environment. The suitability of the data for normal distribution will be evaluated by Shaphiro Wilk Test. For continuous variables with normal distribution, t-test in independent groups will be used to compare two independent group averages; Mann-Whitney U test will be used to compare continuous variables that do not show normal distribution. Statistical significance value will be taken as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Written permission to participate in the study,
* Conscious, oriented and cooperative,
* Speaks and understands Turkish,
* Literate,
* Undergoing TURP,
* No vision problems,
* Patients who or their caregivers have a phone/tablet with the ability to download mobile training

Exclusion Criteria:

* Undergoing TURP for the second time,
* Physically or mentally ill with a physical or mental illness that prevents communication,
* Underwent day surgery,
* Neither they nor their caregivers have a phone/tablet with the ability to download mobile training patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | 10 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).
Anxiety | 10 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Hemodynamic Variables | 10 months
  Hemodynamic Variables Monitoring Form, hemodynamic variables findings of the mobile treatment and control group before and after TURP will be recorded.
Surgical Fear | 10 months
  Surgical Fear Scale: The Turkish validity and reliability study of the scale was conducted by Bağdigen and Karaman Özlü in 2018. The questionnaire, which consists of eight items, has an 11-point Likert structure ranging from 0 (I am not afraid at all) to 10 (I am very afraid). The questionnaire has two subscales indicating the fear of short-term and long-term consequences of surgery. The subscale score is obtained by summing the scores of the four items in the subscales of the questionnaire. The total score of the questionnaire will be obtained by summing the scores of the two subscales, with a minimum score of 0 and a maximum score of 80. The Cronbach alpha coefficient of the scale was found to be 0.89, 0.86 for the short-term outcomes sub-dimension and 0.87 for the long-term outcomes (Bağdiven & Karaman Özlü, 2016).
Education Satisfaction | 10 months
  Education Satisfaction Scale:It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no good at all)-10 (very severe good) to evaluate the level of patient education satisfaction
Urinalysis results | 10 months
  Hemodynamic Variables Monitoring Form, complete urinalysis (density, bacteriuria, etc.) findings of the mobile treatment and control group before and after TURP will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Bozlu, Principal Investigator — Mersin University
Locations (1):
- Tarsus University, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belarmino A, Walsh R, Alshak M, Patel N, Wu R, Hu JC. Feasibility of a Mobile Health Application To Monitor Recovery and Patient-reported Outcomes after Robot-assisted Radical Prostatectomy. Eur Urol Oncol. 2019 Jul;2(4):425-428. doi: 10.1016/j.euo.2018.08.016. Epub 2018 Sep 10. PMID 31277778
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Result] Deniz-Garcia A, Fabelo H, Rodriguez-Almeida AJ, Zamora-Zamorano G, Castro-Fernandez M, Alberiche Ruano MDP, Solvoll T, Granja C, Schopf TR, Callico GM, Soguero-Ruiz C, Wagner AM; WARIFA Consortium. Quality, Usability, and Effectiveness of mHealth Apps and the Role of Artificial Intelligence: Current Scenario and Challenges. J Med Internet Res. 2023 May 4;25:e44030. doi: 10.2196/44030. PMID 37140973
- [Result] Elterman D, Aube-Peterkin M, Evans H, Elmansy H, Meskawi M, Zorn KC, Bhojani N. UPDATE - Canadian Urological Association guideline: Male lower urinary tract symptoms/benign prostatic hyperplasia. Can Urol Assoc J. 2022 Aug;16(8):245-256. doi: 10.5489/cuaj.7906. No abstract available. PMID 35905485